CLINICAL TRIAL: NCT03871998
Title: Short-term Topical Application to Prevent Atopic Dermatitis
Acronym: STOP AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Jonathan Hourihane, Principal Investigator, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STOP AD
Record Dates: First submitted 2019-03-07; First posted 2019-03-12 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Eczema Atopic Dermatitis; Eczema; Eczema, Infantile; Food Allergy
Keywords: Eczema; Atopic dermatitis; Food allergy; Skin barrier; Filaggrin; Natural moisturizing factor; TEWL; Skin microbiome; Prevention; Moisturizer
MeSH Terms: conditions — Eczema; Dermatitis, Atopic; Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Single-centre, randomised, open-label, controlled study to evaluate whether short-term skin barrier protection using a moisturizer from birth to 2 months can prevent the onset of atopic dermatitis and food allergy at 12 months. Assessments of atopic dermatitis will be blinded.
Who Masked: Outcomes Assessor
Masking Description: Research personnel responsible for conducting atopic dermatitis assessments during study follow-up visits will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): Skin barrier protection in the first 2 months of life.
  Interventions: Other: Skin barrier protection in the first 2 months of life
- Control arm (No Intervention): Standard skincare advice. No moisturiser in the first 2 months.

INTERVENTIONS:
Other: Skin barrier protection in the first 2 months of life — Skin barrier protection in the first 2 months of life using a commercially available moisturiser from birth 2 months. Twice daily, whole-body application.
  Arms: Interventional arm

SUMMARY:
This is a randomised, open-label, controlled study designed to investigate the effect of short-term neonatal skin barrier protection using a commercially available moisturiser on the prevention of atopic dermatitis and food allergy in high risk children.

DETAILED DESCRIPTION:
Eczema, also known medically as Atopic Dermatitis (AD) is the most common skin disease of childhood, affecting 20% of Irish children, and is a general term for a group of skin conditions that cause the skin to become dry, red, itchy and inflamed. AD is often the first manifestation of atopic comorbidities including food allergy, asthma and allergic rhinitis. Recently published studies suggest that skin barrier preservation, with topically applied moisturisers in the first year of life, reduces the incidence of AD. Our own data suggests that an earlier window for this skin barrier protection may exist.

This study is a randomised, open-label, controlled study and will investigate the effect of short-term neonatal skin barrier protection on the prevention of AD and food allergy in high risk infants. Infants with at least one parent with a positive history of atopic disease (AD, allergic rhinitis, asthma or food allergy) will be eligible for recruitment.

The first study visit will take place within approximately 4 days of birth in the postnatal wards. At this visit, infants will be randomised to either treatment with skin barrier protection using a commercially available moisturiser or to standard routine skincare with no moisturiser from as soon as possible after birth until 2 months of age. This visit will also involve measurements of neonatal trans-epidermal water loss (TEWL) and natural moisturising factor (NMF) to assess skin barrier function and structure. Skin swabs will also be taken for microbiome and immune biomarker analysis.

Follow-up assessments will take place at 2, 4 and 8 weeks, 6 and 12 months. Each visit will include a physical examination of the infant's skin, including TEWL and NMF measurements, and a questionnaire on infant health, bathing and skincare.

Infant skin swabs will be taken again at 8 weeks and 12 months. A research nurse or doctor, blind to treatment allocation, will administer standardised assessments for the presence (yes/no), extent and severity of AD at 6 and 12 months. Suspected cases of food allergy will be investigated using skin prick testing (SPT) and oral food challenges.

A DNA sample will be taken to test for filaggrin loss-of-function mutations, which are linked to AD risk.

The primary outcome is AD at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy full-term infants, gestational age >36+6 weeks.
* Infant has at least one parent with self-reported atopic dermatitis, food allergy, allergic rhinitis or asthma.
* Not requiring admission to the Neonatal Unit.

Exclusion Criteria:

* No parental history of atopic disease.
* Admission to the Neonatal Unit for issues other than the establishment of normal feeding.
* Being administered oral or parenteral antibiotics.
* Receiving phototherapy for hyperbilirubinaemia.
* Sibling, including twin, already recruited.
* Other serious health issues (e.g. abdominal wall defects, congenital heart disease etc.) or a severe widespread skin condition (e.g. collodion).
* Any condition that would make the use of skin barrier protectant inadvisable or not possible (e.g. ankle talipes or developmental dysplasia of the hip, requiring a Pavlik's harness or casts).
* Participation in any other clinical trial of an investigational medicinal product.

Ages: 0 Days to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 321 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of atopic dermatitis at 12 months. | 12 months
Cumulative incidence of IgE-mediated food allergy at 2 years | 2 years

SECONDARY OUTCOMES:
Longitudinal changes in transepidermal water loss (TEWL) from birth to 12 months | Birth to 12 months
  TEWL measured at birth, 2, 4 and 8 weeks and at 6 and 12 months.
Longitudinal changes in natural moisturising factor (NMF) in the stratum corneum from birth to 12 months. | Birth to 12 months
  NMF measured by Raman spectroscopy at birth, 2, 4 and 8 weeks and at 6 and 12 months.
Microbial diversity and richness of the cheek and antecubital fossa (study subset). | Skin swabs for microbiome analysis will be taken at baseline (0-4 days), 8 weeks and 12 months.
  Microbial community analysis (identification and abundance of a taxonomic units) will be used for the calculations of population diversity and richness indices (rarefaction, Shannon index, abundance-based coverage estimators (ACE), and Chao1) in a subset of study participants (n = 30 per study group).
Changes in skin microbial diversity and richness over the first year of life. | Skin swabs for microbiome analysis will be taken at baseline (0-4 days), 8 weeks and 12 months.
  Comparison of microbial diversity and richness of the cheek and antecubital fossa between baseline, 8 weeks and 12 months (n = 30 per study group).
Comparison of microbial diversity and richness between the intervention and control groups. | Skin swabs for microbiome analysis will be taken at baseline (0-4 days), 8 weeks and 12 months.
  Comparison of microbial diversity and richness of the cheek and antecubital fossa at each timepoint between the intervention (moisturiser) and control (no moisturiser) groups (n = 30 per study group).
Skin biomarker profile analysis of the cheek and antecubital fossa (study subset). | Skin swabs for biomarker analysis will be taken at baseline (0-4 days), 8 weeks and 12 months.
  Cheek and antecubital fossa skin biomarker analysis, including interleukins, chemokines. and antimicrobial peptides (final list to be established) at birth, 8 weeks and 12 months (n = 30 from each study group).
Changes in skin biomarker profile between study over the first year of life. | Skin swabs for biomarker analysis will be taken at baseline (0-4 days), 8 weeks and 12 months.
  Comparison of skin biomarker profiles of the cheek and antecubital fossa between baseline, 8 weeks and 12 months (n = 30 per study group).
Comparison of skin biomarker profiles between the intervention and control groups. | Skin swabs for biomarker analysis will be taken at baseline (0-4 days), 8 weeks and 12 months.
  Comparison of skin biomarker profiles of the cheek and antecubital fossa at each timepoint between the intervention (moisturiser) and control (no moisturiser) groups (n = 30 per group).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan O'B Hourihane, MD, Principal Investigator — Royal College of Surgeons in Ireland
Locations (1):
- Cork University Maternity Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided